CLINICAL TRIAL: NCT06156371
Title: The Effect of Lymphatic Drainage Massage on Interdialytic Weight Gain and Fatigue in Patients Undergoing Hemodialysis
Brief Title: The Effect of Lymphatic Drainage Massage on Interdialytic Weight Gain and Fatigue
Acronym: MLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ezgi ÖNEN EFECAN, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Eonenefecan001
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-01

CONDITIONS: Interdialytic Weight Gain; Fatigue
Keywords: Interdialytic weight gain; Fatigue; Lymphatic drainage; Massage; Hemodialysis
MeSH Terms: conditions — Fatigue | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: prospective, randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Individuals to be sampled will be assigned to groups according to the permutated block randomization method. Block size will be taken as 6. Random numbers will be generated in Excel by a researcher other than the researcher who collected the data, and a suitable number of blocks will be created for the sample. Assignment to groups will be made using the blocks of 6 corresponding to this number in the table. Index cards prepared in accordance with the assignment list will be placed in closed opaque envelopes and serial numbers will be written on them. The envelopes will be kept by a person who does not participate in the study and the assignment order will be learned from this person. The data will be recorded as coded as A, B and C, statistical analyzes will be carried out by the researcher who did not participate in the data collection phase according to this code, and the research report will be written in coded form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lymphatic drainage massage (Experimental): In the lymphatic drainage massage group, a patient will receive a total of 12 treatments, 20 minutes a day, 3 days a week for 4 weeks. Face-to-face manual lymphatic drainage massage will be performed at least 1 hour after the patient starts hemodialysis treatment, according to the morning and afternoon work schedules of the institutions. Manual lymphatic drainage massage will be performed by a certified researcher in accordance with the application steps.
  Interventions: Other: lymphatic drainage massage
- Classic massage (Active Comparator): A patient in the classical massage group will receive a total of 12 treatments, 15 minutes a day, 3 days a week for 4 weeks. The classical face-to-face massage application will be performed at least 1 hour after the patient starts hemodialysis treatment, according to the morning and afternoon work schedules of the institutions.
  Classical massage application will be performed by the researcher. The order of application is upper leg, lower leg and feet. During the application, appropriate methods such as effleurage (stroking), kneading, friction, impact and vibration, which are frequently used in classical massage, will be used. Olive oil will be used as essential oil during application.
  Interventions: Other: classic massage
- Control (No Intervention): No intervention other than the first and last evaluation will be applied to the control group. Patients in this group will continue to receive their usual hemodialysis treatment and care.

INTERVENTIONS:
Other: lymphatic drainage massage — Before the application, the patient will be placed in a supine position and the feet will be elevated to 45 degrees by the researcher. After the infraclavicular lymph node, located at the point where the veins in the neck area meet the thymus gland, is stimulated with a pumping action, lower extremity applications will be started in the form of upper legs, lower legs and feet; By stimulating the inguinal lymph node in the upper leg application, the popliteal lymph node in the lower leg application, and the medial malleolus lymph node in the foot application, the mobility of the lymph fluid in the direction of the stimulated lymph node is used using "stroking, pumping, circular movements or rolling movements" according to the weight characteristic, body type and preference of the patient. will be provided. Finally, passive exercise will be performed 5 times, repeating both legs in flexion and extension positions, and the infraclavicular lymph node will be stimulated.
  Arms: Lymphatic drainage massage
Other: classic massage — The application will be done by the researcher. The order of application is upper leg, lower leg and feet. During the application, appropriate methods such as effleurage (stroking), kneading, friction, impact and vibration will be used. The application will start with efflorescence and end with the same technique. To the upper leg; Starting from the knee to the groin, to the lower leg; The application will be made in the direction of the muscle fibers, starting from the ankle to the knee. Appropriate techniques will be used depending on the characteristics of the application areas, and each technique will be repeated 5-10 times. In the final stage, passive exercise will be performed by moving to the foot and applying flexion and extension to the ankle 5 times. The application will be completed by applying similar applications to the upper and lower legs on the back of the foot and the outer and lower surface of the foot. Olive oil will be used as essential oil during application.
  Arms: Classic massage

SUMMARY:
The aim of this study is to evaluate the effect of lymphatic drainage massage on interdialytic weight gain and fatigue in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
Since there is no similar study in the literature, a preliminary application was made to determine the sample size. According to the inclusion criteria, after reaching a total of 36 people, namely Intervention I = 12, Intervention II = 12 and control group = 12, a power analysis was performed, and the minimum sample size to be taken with 5% type 1 error and 80% power was determined as 60 people. Considering that there might be a 25% loss in the sample, it was decided to include 25 people in the Intervention I group, 25 in the Intervention II group and 25 in the control group, making a total of 75 people, namely Intervention I = 25, Intervention II = 25, Control = 25.36 people. A patient in Intervention 1 (n=25) group will receive a lymphatic drainage massage for 20 minutes a day, 3 days a week, a total of 12 times for 4 weeks. The application will start 1 hour after the patient enters hemodialysis. Before the application, the patient will be placed in a supine position and the researcher will ensure that the feet are elevated to 45 degrees for the application to be effective. In practice, after the infraclavicular lymph node, which is located at the point where the veins in the neck area meet the thymus gland and called the "main terminal" lymph node, is stimulated with a pumping action, lymphatic drainage will be applied to the upper legs, lower legs and feet. A patient in Intervention 2 (n=25) group will receive classical massage on the upper legs, lower legs and feet for 15 minutes a day, 3 days a week, a total of 12 times for 4 weeks. The application will start 1 hour after the patient enters hemodialysis. No intervention other than the first and last evaluation will be applied to the control group. At the end of the study, participants will be given full information, stating that they were not informed about the specific purpose of the study for scientific reasons. The effect of lymphatic drainage massage on interdialysis weight gain and fatigue are the primary outcomes of the study. The effect of lymphatic drainage massage on blood pressure and laboratory findings are secondary outcomes of the study. The results will be collected before and after intervention in the 1st, 2nd, 3rd and 4th weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis at Private Ata Dialysis Center, Private Diamer Dialysis Center, Mersin Nephrology Private Dialysis Center and Private Mersin Dialysis Center between 30.11.2023-30.06.2024 coming for treatment,
* Receiving hemodialysis treatment 3 times a week for at least 6 months,
* The average interdialytic weight gain in the last 3 sessions exceeds 4% of the dry weight,
* Volunteer to participate in the research and
* Individuals who can speak and understand Turkish will be included in the research.

Exclusion Criteria:

* Using insulin,
* Diagnosed with malignant tumor,
* Having deep vein thrombosis and heart failure diagnosed by a physician,
* Those with missing limbs or infected, open wounds in the application areas,
* Pregnant and
* Individuals who are in another complementary treatment program will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Interdialytic weight gain | Change before the application and in the 1st, 2nd, 3rd, and 4th weeks of the application
  In hemodialysis centers, patients' weights are measured and recorded with an electronic scale by the healthcare personnel working in the institution before and after each hemodialysis session. Measurements are made by removing the patients' jackets/coats and shoes. The measurements will be recorded in kilograms by the researcher and weekly interdialytic weight gain will be evaluated.
Fatigue evaluated using the Fatigue Severity Scale | Change before the application and 4th week of the application
  The Turkish validity and reliability of the scale, which was developed by Krupp et al. in 1989, was tested by Armutlu et al. in 2007, and the Cronbach's alpha coefficient was found to be 0.89, and the test-retest reliability was 0.81 (p = 0.719, within 99% confidence interval). The scale, which evaluates individuals' fatigue status in the last month, consists of a total of 9 items and each item is scored between 1-7. "Strongly disagree = 1", "moderately disagree = 2", "somewhat disagree = 3", "neither agree nor disagree = 4", "somewhat agree = 5", "moderately agree = 6", "strongly agree = It is evaluated as 7" points. The total score calculation of the scale is calculated by adding up the scores given to each item to 9.
  It is done by dividing. The lowest score that can be obtained from the scale is 1 and the highest score is 7. A total score of 4 or more from the scale indicates severe fatigue. A higher score indicates increased fatigue.

SECONDARY OUTCOMES:
Blood pressure measurement | Change before the application and in the 1st, 2nd, 3rd, and 4th weeks of the application
  Blood pressure measurements of the patients will be taken before and after the application. A calibrated blood pressure monitor provided by the researcher will be used for all patients during measurements. Blood pressure measurements will be made and recorded at the dialysis center by healthcare personnel who are not involved in the research. The average systolic and diastolic blood pressure values of the patients will be calculated and evaluated weekly.
Evaluation of biochemical findings | Change before the application and 4th week of the application
  With permission from the institutions and patients, previously performed laboratory tests will be evaluated and recorded retrospectively. From laboratory findings, albumin, urea, creatinine, sodium, potassium, calcium, phosphorus and urea clearance will be evaluated.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Turkey, Mersin University, Mersin
  - Mersin Nephrology Private Dialysis Center, Private Ata Dialysis Center, Private Diamer Dialysis Center and Private Mersin Dialysis Center', Yenişehir